CLINICAL TRIAL: NCT00455195
Title: An Open-Label Extension Study of Patients With Late-Onset Pompe Disease Who Were Previously Enrolled in Protocol AGLU02704
Brief Title: Late-Onset Treatment Study Extension Protocol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGLU03206; 2006-003644-31 (EudraCT Number)
Expanded Access: NCT00520143 (Approved for marketing)
Record Dates: First submitted 2007-03-30; First posted 2007-04-03 (Estimated); Results first posted 2012-01-05 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-02

CONDITIONS: Pompe Disease (Late-Onset); Glycogen Storage Disease Type II (GSD-II); Glycogenesis Type II; Acid Maltase Deficiency (AMD)
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alglucosidase Alfa/Alglucosidase Alfa (Experimental): Participants who received alglucosidase alfa during the double-blind study and, if they completed the double-blind study, continued that treatment during the extension study. Participants received an intravenous (IV) infusion of 20 mg/kg of alglucosidase alfa every other week (qow) until their participation in both the AGLU02704 (NCT00158600) and AGLU03206 studies combined equaled a minimum of 104 weeks.
  Interventions: Biological: alglucosidase alfa
- Placebo/Alglucosidase Alfa (Experimental): Participants given placebo during the double-blind study, completed the double-blind study (study AGLU02704, NCT00158600), and qualified to continue into the extension study on alglucosidase alfa. Participants received an intravenous (IV) infusion of 20 mg/kg of alglucosidase alfa every other week (qow) for up to 52 weeks. Only the alglucosidase alfa treatment experience is included in this extension study.
  Interventions: Biological: alglucosidase alfa

INTERVENTIONS:
Biological: alglucosidase alfa — IV infusion of 20 mg/kg; every other week (qow)
  Other Names: Myozyme; Lumizyme

SUMMARY:
Pompe disease (also known as glycogen storage disease Type II) is caused by a deficiency of a critical enzyme in the body called acid alpha-glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In patients with Pompe disease, an excessive amount of glycogen accumulates and is stored in various tissues, especially heart and skeletal muscle, which prevents their normal function. The objective of this extension study is to assess the long-term safety and efficacy of alglucosidase alfa treatment in patients with Late-Onset Pompe Disease who were previously treated under the placebo-controlled, double-blind study AGLU02704 (NCT00158600).

ELIGIBILITY:
Inclusion Criteria:

* Patient must have completed protocol AGLU02704 (NCT00158600)
* Patient must provide signed, informed consent prior to performing any study-related procedures
* Patient (and patient's legal guardian if patient is under 18 years of age) must have the ability to comply with the clinical protocol
* A female patient of childbearing potential must have a negative pregnancy test at Baseline. (note: all female patients of childbearing potential and sexually mature males must use a medically accepted method of contraception throughout the study.)

Exclusion Criteria:

* The patient has a medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, would preclude treatment with alglucosidase alfa.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (31):
- United States (26):
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Beverly Hills, California
  - San Diego, California
  - Washington D.C., District of Columbia
  - Coral Springs, Florida
  - Gainesville, Florida
  - Sarasota, Florida
  - Chicago, Illinois
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Omaha, Nebraska
  - New York, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Greenville, South Carolina
  - Dallas, Texas
  - San Antonio, Texas
  - Seattle, Washington
  - Green Bay, Wisconsin
- Westmead, Australia
- Canada (2):
  - Calgary, Alberta
  - Sherbrooke, Quebec
- Paris, France
- Rotterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 81 of the 90 participants enrolled in the double-blind placebo controlled AGLU02704 (NCT00158600) study continued on to the open-label extension study AGLU03206.
Groups:
- Alglucosidase Alfa/Alglucosidase Alfa: Participants who received alglucosidase alfa during the double-blind study AGLU02704 (NCT00158600) and, if they completed the double blind study, continued alglucosidase alfa in the extension study. Both study experiences on alglucosidase alfa are represented within AGLU03206.
- Placebo/Alglucosidase Alfa: Participants who received placebo during the double-blind study AGLU02704 (NCT00158600), completed the double-blind study, and started alglucosidase alfa in the extension study. Only participants' experience on alglucosidase alfa in the extension study is represented.
Period: Double-blind Study AGLU02704
Arm/Group | Alglucosidase Alfa/Alglucosidase Alfa | Placebo/Alglucosidase Alfa
Started | 60 (Patients randomized to alglucosidase alfa treatment group in AGLU02704 (NCT00158600).) | 30 (See study AGLU02704 (NCT00158600) for results while on placebo.)
Completed | 55 | 26
Not Completed | 5 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Unable to commit time to study | 0 | 1
Period: Extension Study AGLU03206
Arm/Group | Alglucosidase Alfa/Alglucosidase Alfa | Placebo/Alglucosidase Alfa
Started | 55 | 26 (These 26 participants completed placebo double-blind treatment in the AGLU02704 (NCT00158600) study.)
Completed | 55 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alglucosidase Alfa/Alglucosidase Alfa | Placebo/Alglucosidase Alfa | Total
Number analyzed (Participants) | 60 | 26 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at first infusion of alglucosidase alfa. The Alglucosidase Alfa/Alglucosidase Alfa treatment arm includes participants' study experience in the double-blind study (AGLU02704 (NCT00158600)) and the extension study (AGLU03206 (NCT00455195) hence 60 participants are represented. The Placebo/Alglucosidase Alfa treatment arm includes participants' study experience on Alglucosidase Alfa in the extension study (AGLU03206) hence 26 participants are represented.
  years | 45.3 (12.37) | 46.8 (8.62) | 45.73 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants] — The Alglucosidase Alfa/Alglucosidase Alfa treatment arm includes participants' study experience in the double-blind study (AGLU02704 (NCT00158600)) and the extension study (AGLU03206 (NCT00455195) hence 60 participants are represented. The Placebo/Alglucosidase Alfa treatment arm includes participants' study experience on Alglucosidase Alfa in the extension study (AGLU03206) hence 26 participants are represented.
  Participants
    Female | 26 | 15 | 41
    Male | 34 | 11 | 45
Race/Ethnicity, Customized [Number; unit: participants] — The Alglucosidase Alfa/Alglucosidase Alfa treatment arm includes participants' study experience in the double-blind study (AGLU02704 (NCT00158600)) and the extension study (AGLU03206 (NCT00455195) hence 60 participants are represented. The Placebo/Alglucosidase Alfa treatment arm includes participants' study experience on Alglucosidase Alfa in the extension study (AGLU03206) hence 26 participants are represented.
  participants
    Hispanic | 1 | 1 | 2
    Asian | 1 | 0 | 1
    Black or African American | 0 | 0 | 0
    White | 57 | 24 | 81
    Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Summary of Participants Reporting Treatment-Emergent Adverse Events For Participants Treated With Alglucosidase Alfa During Study AGLU02704 (NCT00158600)
Description: The numbers of participants who experienced Adverse Events (AEs), Serious Adverse Events (SAEs), treatment-related AEs, and Infusion Associated Reactions (IARs). Summary is based on treatment-emergent AEs (TEAEs), defined as AEs that occurred following the initiation of study treatment with alglucosidase alfa.
  Participants with long-term exposure to alglucosidase alfa (those from the Alglucosidase Alfa/Alglucosidase Alfa treatment group) are included. Time frames are stated from the start of the double-blind study AGLU02704 (NCT00158600).
Time Frame: Week 0 to 2.5 years
Population: The safety population includes all participants randomized to alglucosidase alfa treatment in AGLU02704 (NCT00158600) who received at least one infusion of alglucosidase alfa.
Measure: Number; unit: participants
Arm/Group | Alglucosidase Alfa/Alglucosidase Alfa
Number analyzed (Participants) | 60
participants
  Participants with any AEs | 60
  Participants with Treatment-Related AEs | 37
  Participants with Infusion-Associated Reactions | 21
  Participants with Serious AEs | 15
  Participants with Severe AEs | 16
  Participants- Discontinued Due to AEs (incl death) | 3
  Participants Who Died | 1

2. Secondary Outcome: Baseline Values (Week 0) for Percent Predicted Proximal Muscle Strength of the Lower Limbs as Measured by Quantitative Muscle Testing (QMT) For Participants Treated With Alglucosidase Alfa During Study AGLU02704 (NCT00158600)
Description: Quantitative muscle testing (QMT) is a standardized system to measure muscle force production during maximal voluntary isometric contraction. QMT data were collected directly from sensors into laptop computers. Predicted normal values for QMT are based on a formula using sex, age and body mass index of a person, and are an estimate of healthy muscle force. Percent of predicted QMT = (observed value)/(predicted value) * 100%. The QMT Leg Score is the average of the bilateral means for percent predicted knee flexors and extensors. A value of 100% indicates 'normal' muscle strength.
Time Frame: Week 0
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent of predicted QMT
Arm/Group | Alglucosidase Alfa/Alglucosidase Alfa
Number analyzed (Participants) | 60
percent of predicted QMT | 37.7 (18.88)

3. Primary Outcome: Baseline Values (Week 0) of Functional Endurance as Measured by Six-Minute Walk Test (6MWT) For Participants Treated With Alglucosidase Alfa During Study AGLU02704 (NCT00158600)
Description: Six-Minute Walk Test (6MWT) measures the distance walked (in meters) in 6 minutes. A longer distance indicates greater endurance. Time frames are stated from the start of the double-blind study AGLU02704 (NCT00158600).
Time Frame: Week 0
Population: Intent-to-treat population.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Alglucosidase Alfa/Alglucosidase Alfa
Number analyzed (Participants) | 60
meters | 332.2 (126.69)

4. Primary Outcome: Change From Baseline (Week 0) in the Six-Minute Walk Test (6MWT) at Week 104 For Participants Treated With Alglucosidase Alfa During Study AGLU02704 (NCT00158600)
Description: Six-Minute Walk Test (6MWT) measures the distance walked (in meters) in 6 minutes. A longer distance indicates greater endurance. Time frames are stated from the start of the double-blind study AGLU02704 (NCT00158600). Change is calculated as the value minus the baseline value.
Time Frame: Week 0, Week 104
Population: Intent-to-treat population of participants who had both baseline (Week 0) and Week 104 data.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Alglucosidase Alfa/Alglucosidase Alfa
Number analyzed (Participants) | 53
meters | 21.3 (78.02)

5. Secondary Outcome: Change From Baseline (Week 0) for Percent Predicted Proximal Muscle Strength of the Lower Limbs as Measured by Quantitative Muscle Testing (QMT) at Week 104 For Participants Treated With Alglucosidase Alfa During Study AGLU02704 (NCT00158600)
Description: as for outcome 2
Time Frame: Week 0, Week 104
Population: Intent-to-treat population of participants who had both baseline (Week 0) and Week 104 data.
Measure: Mean (Standard Deviation); unit: percent of predicted QMT
Arm/Group | Alglucosidase Alfa/Alglucosidase Alfa
Number analyzed (Participants) | 53
percent of predicted QMT | 2.1 (11.06)

6. Primary Outcome: Baseline Values (Week 0) for Percent Predicted Forced Vital Capacity (FVC) For Participants Treated With Alglucosidase Alfa During Study AGLU02704 (NCT00158600)
Description: Forced vital capacity (FVC) is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC is the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted forced vital capacity is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FVC = (observed value)/(predicted value) * 100%. Time frames are stated from the start of the double-blind study AGLU02704 (NCT00158600).
Time Frame: Week 0
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent of predicted FVC
Arm/Group | Alglucosidase Alfa/Alglucosidase Alfa
Number analyzed (Participants) | 60
percent of predicted FVC | 55.4 (14.44)

7. Primary Outcome: Change From Baseline (Week 0) in the Percent Predicted Forced Vital Capacity (FVC) at Week 104 For Participants Treated With Alglucosidase Alfa During Study AGLU02704 (NCT00158600)
Description: Forced vital capacity (FVC) is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC is the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Predicted forced vital capacity is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FVC = (observed value)/(predicted value) * 100%. Time frames are stated from the start of the double-blind study AGLU02704 (NCT00158600). Change is calculated as the value minus the baseline value.
Time Frame: Week 0, Week 104
Population: Intent-to-treat population of participants who had both baseline (Week 0) and Week 104 data.
Measure: Mean (Standard Deviation); unit: percent of predicted FVC
Arm/Group | Alglucosidase Alfa/Alglucosidase Alfa
Number analyzed (Participants) | 53
percent of predicted FVC | 0.8 (6.68)

8. Secondary Outcome: Baseline Values (Week 0) for Quality of Life Related to Physical Component Score (PCS) as Measured by the Medical Outcomes Study (MOS) Short Form-36 Health Survey For Participants Treated With Alglucosidase Alfa During Study AGLU02704 (NCT00158600)
Description: The Medical Outcomes Study Short Form (MOS SF)-36 questionnaire consists of 36 items grouped into 8 domains designed to assess generic health-related quality of life in healthy and ill adult populations. Physical Component Score reports the four domains of physical functioning, role-physical, bodily pain, and general health and are standardized as Z-scores (scale of 0-100). Higher scores are associated with better quality of life. Time frames are stated from the start of the double-blind study AGLU02704 (NCT00158600).
Time Frame: Week 0
Population: Intent-to-treat population of participants with valid baseline (Week 0) PCS surveys.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alglucosidase Alfa/Alglucosidase Alfa
Number analyzed (Participants) | 58
units on a scale | 34.33 (8.934)

9. Secondary Outcome: Change From Baseline in Quality of Life Related to Physical Component Score (PCS) as Measured by the Medical Outcomes Study (MOS) Short Form-36 Health Survey For Participants Treated With Alglucosidase Alfa During Study AGLU02704 (NCT00158600)
Description: The Medical Outcomes Study Short Form (MOS SF)-36 questionnaire consists of 36 items grouped into 8 domains designed to assess generic health-related quality of life in healthy and ill adult populations. Physical Component Score reports the four domains of physical functioning, role-physical, bodily pain, and general health and is standardized as Z-scores (scale of 0-100). Higher scores are associated with better quality of life. Change is calculated as the value minus the baseline value. Time frames are stated from the start of the double-blind study AGLU02704 (NCT00158600).
Time Frame: Week 0 , Week 104
Population: Intent-to-treat population of participants who had valid baseline (Week 0) and Week 104 data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alglucosidase Alfa/Alglucosidase Alfa
Number analyzed (Participants) | 49
units on a scale | 0.64 (7.618) [-1.6 to 2.8]

ADVERSE EVENTS:
Time Frame: Adverse events for the Alglucosidase Alfa/Alglucosidase Alfa group cover up to 2.5 years (Week 0 to 2.5 years), and for the Placebo/Alglucosidase Alfa group cover up to 1.0 year (Week 78 to 2.5 years).
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables. Events are listed independent of relationship to treatment reported.
Groups:
- Placebo/Alglucosidase Alfa: Participants who received placebo during the double-blind study AGLU02704 (NCT00158600) and, if they completed the double-blind study, started alglucosidase alfa in the extension study. Only participants' experience on alglucosidase alfa in the extension study is represented.
- Overall: The combined alglucosidase alfa treatment experience from the two treatment groups.
Arm/Group | Alglucosidase Alfa/Alglucosidase Alfa | Placebo/Alglucosidase Alfa | Overall
Serious Adverse Events (participants affected / at risk) | 15/60 | 2/26 | 17/86
Other Adverse Events (participants affected / at risk) | 60/60 | 25/26 | 85/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alglucosidase Alfa/Alglucosidase Alfa (N=60) | Placebo/Alglucosidase Alfa (N=26) | Overall (N=86)
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Brain stem ischaemia (Nervous system disorders) | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Aneurysm (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alglucosidase Alfa/Alglucosidase Alfa (N=60) | Placebo/Alglucosidase Alfa (N=26) | Overall (N=86)
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 5 | 0 | 5
Macrocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Atrial hypertrophy (Cardiac disorders) | 1 | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 3 | 0 | 3
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0 | 2
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 1
Ventricular dysfunction (Cardiac disorders) | 0 | 1 | 1
Ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 1
Auricular swelling (Ear and labyrinth disorders) | 1 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 1
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 5 | 0 | 5
Ear pain (Ear and labyrinth disorders) | 3 | 0 | 3
Hypoacusis (Ear and labyrinth disorders) | 23 | 3 | 26
Presbyacusis (Ear and labyrinth disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 5 | 0 | 5
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 1
Altered visual depth perception (Eye disorders) | 1 | 0 | 1
Asthenopia (Eye disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 4 | 1 | 5
Conjunctivitis (Eye disorders) | 1 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 1
Eye irritation (Eye disorders) | 1 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0 | 1
Eyelid ptosis (Eye disorders) | 1 | 0 | 1
Keratoconjunctivitis sicca (Eye disorders) | 0 | 1 | 1
Photophobia (Eye disorders) | 1 | 0 | 1
Pinguecula (Eye disorders) | 1 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 4 | 0 | 4
Visual acuity reduced (Eye disorders) | 1 | 0 | 1
Visual disturbance (Eye disorders) | 1 | 0 | 1
Vitreous floaters (Eye disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 2
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 5
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 6 | 1 | 7
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 1
Anorectal disorder (Gastrointestinal disorders) | 1 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Bowel sounds abnormal (Gastrointestinal disorders) | 0 | 1 | 1
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 7 | 0 | 7
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 20 | 2 | 22
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 7 | 0 | 7
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0 | 2
Food poisoning (Gastrointestinal disorders) | 2 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 2
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 2 | 1 | 3
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 15 | 2 | 17
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 1
Oral pruritus (Gastrointestinal disorders) | 1 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 3 | 0 | 3
Swollen tongue (Gastrointestinal disorders) | 2 | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 14 | 2 | 16
Adverse drug reaction (General disorders) | 1 | 0 | 1
Application site vesicles (General disorders) | 1 | 0 | 1
Asthenia (General disorders) | 4 | 0 | 4
Axillary pain (General disorders) | 1 | 0 | 1
Catheter related complication (General disorders) | 1 | 0 | 1
Catheter site pain (General disorders) | 2 | 0 | 2
Chest discomfort (General disorders) | 7 | 0 | 7
Chest pain (General disorders) | 6 | 2 | 8
Chills (General disorders) | 4 | 1 | 5
Disease progression (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 13 | 4 | 17
Feeling abnormal (General disorders) | 1 | 0 | 1
Feeling cold (General disorders) | 2 | 0 | 2
Feeling hot (General disorders) | 3 | 0 | 3
Gait disturbance (General disorders) | 1 | 0 | 1
Influenza like illness (General disorders) | 2 | 0 | 2
Infusion site bruising (General disorders) | 1 | 0 | 1
Infusion site pain (General disorders) | 2 | 0 | 2
Infusion site paraesthesia (General disorders) | 1 | 0 | 1
Infusion site reaction (General disorders) | 7 | 0 | 7
Injection site pain (General disorders) | 1 | 0 | 1
Injection site phlebitis (General disorders) | 1 | 0 | 1
Local swelling (General disorders) | 2 | 0 | 2
Malaise (General disorders) | 3 | 0 | 3
Nodule (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 13 | 1 | 14
Pain (General disorders) | 6 | 0 | 6
Pitting oedema (General disorders) | 1 | 0 | 1
Puncture site haemorrhage (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 12 | 2 | 14
Thirst (General disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 1 | 3
Seasonal allergy (Immune system disorders) | 1 | 0 | 1
Acute tonsillitis (Infections and infestations) | 2 | 0 | 2
Bronchiolitis (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 0 | 3
Bronchitis acute (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Cystitis (Infections and infestations) | 2 | 0 | 2
Dermatophytosis (Infections and infestations) | 1 | 0 | 1
Ear infection (Infections and infestations) | 2 | 0 | 2
Eye infection (Infections and infestations) | 1 | 0 | 1
Folliculitis (Infections and infestations) | 2 | 0 | 2
Fungal infection (Infections and infestations) | 2 | 0 | 2
Fungal skin infection (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 8 | 0 | 8
Gastroenteritis viral (Infections and infestations) | 4 | 0 | 4
Gingival infection (Infections and infestations) | 1 | 0 | 1
Herpes simplex (Infections and infestations) | 4 | 1 | 5
Herpes virus infection (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 8 | 3 | 11
Kidney infection (Infections and infestations) | 1 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Mucosal infection (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 29 | 8 | 37
Otitis media (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 3 | 1 | 4
Rhinitis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 9 | 3 | 12
Tinea pedis (Infections and infestations) | 2 | 0 | 2
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 1
Tooth infection (Infections and infestations) | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 20 | 6 | 26
Urinary tract infection (Infections and infestations) | 5 | 2 | 7
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 1
Vaginal infection (Infections and infestations) | 1 | 1 | 2
Viral infection (Infections and infestations) | 2 | 0 | 2
Wound infection (Infections and infestations) | 1 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 9 | 1 | 10
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 39 | 13 | 52
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 4 | 0 | 4
Injury corneal (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 6 | 2 | 8
Neck injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 9 | 1 | 10
Radial nerve injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0 | 2
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 5 | 0 | 5
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0 | 2
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Blood creatine increased (Investigations) | 1 | 0 | 1
Blood folate decreased (Investigations) | 1 | 0 | 1
Blood glucose increased (Investigations) | 1 | 2 | 3
Blood pressure increased (Investigations) | 3 | 0 | 3
Blood uric acid increased (Investigations) | 1 | 0 | 1
Blood urine present (Investigations) | 1 | 0 | 1
Body temperature increased (Investigations) | 1 | 0 | 1
Carbon dioxide increased (Investigations) | 1 | 1 | 2
Crystal urine present (Investigations) | 1 | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 1 | 0 | 1
Electrocardiogram T wave amplitude decreased (Investigations) | 1 | 0 | 1
Electrocardiogram abnormal (Investigations) | 1 | 0 | 1
Fungus urine test positive (Investigations) | 1 | 0 | 1
Glucose urine present (Investigations) | 1 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1 | 1
Neutrophil count increased (Investigations) | 1 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 1
Protein urine present (Investigations) | 3 | 0 | 3
Specific gravity urine increased (Investigations) | 1 | 0 | 1
Tandem gait test abnormal (Investigations) | 1 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 1 | 1
Urine ketone body present (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 2 | 1 | 3
White blood cell count increased (Investigations) | 1 | 0 | 1
White blood cells urine positive (Investigations) | 1 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 4 | 29
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 6 | 25
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Buttock pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 5 | 22
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 6 | 0 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 | 2 | 13
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 7
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 4 | 14
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 8 | 0 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 3 | 19
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 1 | 10
Nose deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 2 | 25
Senile ankylosing vertebral hyperostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Areflexia (Nervous system disorders) | 5 | 2 | 7
Balance disorder (Nervous system disorders) | 3 | 0 | 3
Burning sensation (Nervous system disorders) | 2 | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 16 | 3 | 19
Dizziness postural (Nervous system disorders) | 2 | 0 | 2
Facial palsy (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 31 | 6 | 37
Hyperreflexia (Nervous system disorders) | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 0 | 3
Hyporeflexia (Nervous system disorders) | 3 | 0 | 3
Intercostal neuralgia (Nervous system disorders) | 1 | 0 | 1
Lethargy (Nervous system disorders) | 2 | 1 | 3
Loss of consciousness (Nervous system disorders) | 2 | 0 | 2
Migraine (Nervous system disorders) | 4 | 0 | 4
Nerve compression (Nervous system disorders) | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 7 | 0 | 7
Sciatica (Nervous system disorders) | 1 | 0 | 1
Sensory disturbance (Nervous system disorders) | 1 | 1 | 2
Sinus headache (Nervous system disorders) | 1 | 1 | 2
Somnolence (Nervous system disorders) | 4 | 0 | 4
Syncope vasovagal (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 4 | 1 | 5
Anger (Psychiatric disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 0 | 3
Depression (Psychiatric disorders) | 2 | 0 | 2
Insomnia (Psychiatric disorders) | 9 | 0 | 9
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 1
Stress (Psychiatric disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 2
Haematuria (Renal and urinary disorders) | 3 | 1 | 4
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 3 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 0 | 2
Pyuria (Renal and urinary disorders) | 1 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1 | 1
Urge incontinence (Renal and urinary disorders) | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 1 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 1
Breast swelling (Reproductive system and breast disorders) | 1 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 2
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1
Menstrual discomfort (Reproductive system and breast disorders) | 1 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 2 | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 1 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 8
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 3 | 17
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 1 | 7
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 3 | 11
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 9 | 1 | 10
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 5 | 0 | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 0 | 4
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin inflammation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 7 | 1 | 8
Urticaria contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Aneurysm (Vascular disorders) | 1 | 0 | 1
Cardiovascular insufficiency (Vascular disorders) | 1 | 0 | 1
Diastolic hypotension (Vascular disorders) | 1 | 0 | 1
Flushing (Vascular disorders) | 3 | 1 | 4
Haematoma (Vascular disorders) | 2 | 0 | 2
Hot flush (Vascular disorders) | 2 | 0 | 2
Hypertension (Vascular disorders) | 5 | 0 | 5
Hypotension (Vascular disorders) | 2 | 1 | 3
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 1
Vasoconstriction (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.